CLINICAL TRIAL: NCT02187562
Title: Effect of Steady State Meloxicam 15 mg/Day on Low Dose Aspirin (100 mg/Day) Induced Inhibition of Platelet Aggregation and Thromboxane Synthesis in Healthy Males and Females. An Open, Randomised, Two-way Crossover Study.
Brief Title: Effect of Steady State Meloxicam on Low Dose Aspirin Induced Inhibition of Platelet Aggregation and Thromboxane Synthesis in Healthy Males and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.255
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam; Aspirin

ARMS (2):
- Meloxicam/Aspirin (Experimental): Meloxicam days 1-10 / Aspirin days 5-10
  Interventions: Drug: Meloxicam; Drug: Aspirin
- Aspirin (Active Comparator): Aspirin 2 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Meloxicam
  Arms: Meloxicam/Aspirin
Drug: Aspirin

SUMMARY:
The objective of this study was to investigate the influence of meloxicam on low dose aspirin induced inhibition of platelet aggregation and thromboxane B2, when meloxicam is given before aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <= 60 years
* The Body Mass Index (BMI) ≥ 18.5 kg/m2 (square meters) and ≤ 29.9 kg/m2.
* Laboratory values within a clinical normal range

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, in particular aspirin containing drugs(< 14 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 1 months prior to administration (at least 10 times the relevant elimination half-life) or during trial)
* Having had prescription medication 2 weeks prior to study drug administration or over the counter medication 1 week prior to study drug administration (at least 10 times the relevant elimination half-life)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 grams (g)/day)
* Drug abuse
* Blood donation or loss > 400 mL (< 1 month prior to administration or during the trial)
* Excessive physical activities (< 5 days prior to administration or during the trial)
* Any ECG value outside of the reference range of clinical relevance including, but not limited to QTcB > 480 ms or QRS interval > 110 ms
* History of any familial bleeding disorder
* History of haemorrhagic diatheses
* History of gastrointestinal ulcer, perforation or bleeding
* History of bronchial asthma
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (e.g. sterilisation, intrauterine device (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ovarian hormone substitution and oral contraception have to be continued during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2002-07; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Arachidonic acid induced platelet aggregation | up to day 11 (treatment 1), up to day 3 (treatment 2)

SECONDARY OUTCOMES:
Collagen-induced Platelet Aggregation | up to day 11 (treatment 1), up to day 3 (treatment 2)
Adenosine diphosphate (ADP) Induced Platelet Aggregation | up to day 11 (treatment 1), up to day 3 (treatment 2)
Serum Thromboxane B2 production | up to day 11 (treatment 1), up to day 3 (treatment 2)
Number of patients with adverse events | up to 6 weeks
Number of patients with abnormal changes in laboratory parameters | up to day 11 (treatment 1), up to day 3 (treatment 2)
Number of patients with abnormal changes in 12-lead electrocardiogram (ECG) | Screening, 24 hours after the last Aspirin intake
Number of patients with clinically significant changes in vital signs | Screening, 24 hours after the last Aspirin intake
Assessment of tolerability on a 4-point scale | 24 hours after the last Aspirin intake